CLINICAL TRIAL: NCT03042962
Title: Brain Networks in Dystonia
Status: Recruiting | Type: Observational
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Kristina Simonyan, Professor of Otolaryngology - Head and Neck Surgery, Massachusetts Eye and Ear Infirmary
Other Study IDs: 2019P001183; R01DE030464 (NIH)
Record Dates: First submitted 2017-01-31; First posted 2017-02-03 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Spasmodic Dysphonia; Singer's Dystonia; Writer's Cramp; Musician's Focal Hand Dystonia; Craniofacial Dystonia; Blepharospasm Oromandibular Dystonia
Keywords: dystonia; imaging; genetics
MeSH Terms: conditions — Dysphonia; Dystonic Disorders; Meige Syndrome; Dystonia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples will be collected, the DNA will be extracted and banked for genetic studies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with dystonia and their unaffected relatives: Patients with dystonia and their unaffected blood relatives will undergo MRI of the brain and blood draw.
  Interventions: Other: MRI; Procedure: Blood draw
- Healthy volunteers: Healthy subjects without any neurological, psychiatric or otolaryngological problems will undergo MRI of the brain and blood draw.
  Interventions: Other: MRI; Procedure: Blood draw

INTERVENTIONS:
Other: MRI — Functional and structural MRI of the brain will be conducted to identify disorder specific neural markers
Procedure: Blood draw — Blood samples will be collected, the DNA will be extracted and banked for genetic studies

SUMMARY:
To date, there is only limited knowledge about the distinct neural abnormalities that lead to the development of different forms of focal dystonia. The goal of this study is to dissect the pathophysiological mechanisms underlying this clinical phenomenon using multi-level brain network analysis in patients with focal dystonia.

DETAILED DESCRIPTION:
Among the many causes of craniofacial disease are focal dystonias such as blepharospasm (BSP) and oromandibular dystonia (OMD), affecting the eyes and jaw, respectively, as well as Meige Syndrome, which combines features of both. Craniofacial dystonias are poorly understood and have limited treatment options. The investigators hypothesize that craniofacial dystonia (CFD) may be caused by both rare and common genetic variants. To identify neural correlates of different genetic causes of CFD, the investigators will perform structural and functional whole-brain imaging and examine the organization of the neural network in these patients compared to healthy individuals and their unaffected blood relatives.

ELIGIBILITY:
Inclusion Criteria:

* Patients will have clinically documented focal dystonia
* Unaffected relatives of patients with focal dystonia
* Healthy controls will be healthy volunteers with a negative history of neurological, laryngeal or psychiatric problems
* Age from 21 to 80 years.
* Native English speakers.
* Right-handedness (based on Edinburgh Handedness Inventory).

Exclusion Criteria:

* Subjects who are incapable of giving an informed consent.
* Pregnant or breastfeeding women until a time when they are no longer pregnant or breastfeeding. All women of childbearing potential will have a urine pregnancy test performed, which must be negative for participation in the imaging studies.
* Subjects with past or present medical history of (a) neurological problems, such as stroke, movement disorders (other than dystonia in the patient groups), brain tumors, traumatic brain injury with loss of consciousness, ataxias, myopathies, myasthenia gravis, demyelinating diseases, alcoholism, drug depend-ence; (b) psychiatric problems, such as schizophrenia, major and/or bipolar depression, obsessive-compulsive disorder; (c) laryngeal problems, such as vocal fold paralysis, paresis, vocal fold nodules and polyps, carcinoma, chronic laryngitis.
* Patients who are not symptomatic due to treatment with botulinum toxin injections into the laryngeal muscles. The duration of positive effects of botulinum toxin vary from patient to patient but lasts on average for 3-4 months. All patients will be evaluated to ensure that they are fully symptomatic prior to entering the study.
* Patients with other forms of dystonia.
* Patients who have dystonia symptoms at rest in order to avoid the potential confound of dystonic spasms occurring during the scanning.
* To avoid the possibility of confounding effects of drugs acting upon the central nervous system, all study participants will be questioned about any prescribed or over-the-counter medications as part of their initial intake screening. Those patients who receive medication(s) affecting the central nervous system will be excluded from the study.
* The patients will be asked whether they have undergone any head, neck, or hand surgeries, which resulted in changes in regional anatomy or innervation. Because brain, hand and laryngeal surgery may potentially lead to the brain structure and function re-organization, all patients with history of brain, hand and/or laryngeal surgery will be excluded from the study.
* Subjects who have tattoos, ferromagnetic objects in their bodies (e.g., implanted stimulators, surgical clips, prosthesis, artificial heart valve, etc.) that cannot be removed for the purpose of study participation.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with focal dystonia, thier unaffected blood relatives, and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 141 (Estimated)
Dates: Start 2015-08-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of brain structural and functional changes | 5 years
  Identify changes in brain activity and gray and white matter in patients with dystonia vs. unaffected relatives vs. healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Simonyan, MD, PhD, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Battistella G, Termsarasab P, Ramdhani RA, Fuertinger S, Simonyan K. Isolated Focal Dystonia as a Disorder of Large-Scale Functional Networks. Cereb Cortex. 2017 Feb 1;27(2):1203-1215. doi: 10.1093/cercor/bhv313. PMID 26679193
- [Result] Fuertinger S, Simonyan K. Stability of Network Communities as a Function of Task Complexity. J Cogn Neurosci. 2016 Dec;28(12):2030-2043. doi: 10.1162/jocn_a_01026. Epub 2016 Aug 30. PMID 27575646
- [Result] Rittiner JE, Caffall ZF, Hernandez-Martinez R, Sanderson SM, Pearson JL, Tsukayama KK, Liu AY, Xiao C, Tracy S, Shipman MK, Hickey P, Johnson J, Scott B, Stacy M, Saunders-Pullman R, Bressman S, Simonyan K, Sharma N, Ozelius LJ, Cirulli ET, Calakos N. Functional Genomic Analyses of Mendelian and Sporadic Disease Identify Impaired eIF2alpha Signaling as a Generalizable Mechanism for Dystonia. Neuron. 2016 Dec 21;92(6):1238-1251. doi: 10.1016/j.neuron.2016.11.012. Epub 2016 Dec 8. PMID 27939583
- [Result] Fuertinger S, Simonyan K. Connectome-Wide Phenotypical and Genotypical Associations in Focal Dystonia. J Neurosci. 2017 Aug 2;37(31):7438-7449. doi: 10.1523/JNEUROSCI.0384-17.2017. Epub 2017 Jul 3. PMID 28674168
- [Result] Farouk R, Duthie GS, Pryde A, Bartolo DC. Abnormal transient internal sphincter relaxation in idiopathic pruritus ani: physiological evidence from ambulatory monitoring. Br J Surg. 1994 Apr;81(4):603-6. doi: 10.1002/bjs.1800810442. PMID 8205448
- [Result] [Comparison of pregnancies issued from frozen embryo transfers and pregnancies issued from fresh embryo transfers in fertilization in vitro. FIVNAT]. Contracept Fertil Sex. 1994 May;22(5):287-91. French. PMID 8032380
- [Result] Rosenthal DN, Friedman AH, Kleinman CS, Kopf GS, Rosenfeld LE, Hellenbrand WE. Thromboembolic complications after Fontan operations. Circulation. 1995 Nov 1;92(9 Suppl):II287-93. doi: 10.1161/01.cir.92.9.287. PMID 7586425
- [Result] Hollander E, Toth C. [Severe life threatening metabolic alkalosis]. Orv Hetil. 1980 Feb 17;121(7):391-6. No abstract available. Hungarian. PMID 7375103
- [Result] Kleber FX. Socioeconomic aspects of ACE inhibition in the secondary prevention in cardiovascular diseases. Am J Hypertens. 1994 Sep;7(9 Pt 2):112S-116S. doi: 10.1093/ajh/7.9.112s. PMID 7818836
- [Result] Friederichs H. [Physicians and experts competence law. Indications on the latest legal decisions]. Fortschr Med. 1981 Apr 9;99(14):516. No abstract available. German. PMID 7274927
- [Result] van Niekerk FW, Miller VJ. Diet and dentures. J Dent Assoc S Afr. 1983 Sep;38(9):569, 572. No abstract available. PMID 6581586
- [Result] Stewart P, Calder AA. Cervical ripening. Br J Obstet Gynaecol. 1981 Oct;88(10):1071-2. No abstract available. PMID 6945119
- [Result] Hirst GK. Presentation of Academy Medal to Edwin D. Kilbourne, M.D. Bull N Y Acad Med. 1983 Sep;59(7):626-31. No abstract available. PMID 6354324
- [Result] St-Arnaud R, Walker P, Kelly PA, Labrie F. Rat ovarian epidermal growth factor receptors: characterization and hormonal regulation. Mol Cell Endocrinol. 1983 Jul;31(1):43-52. doi: 10.1016/0303-7207(83)90029-1. PMID 6309584
- [Result] Steendijk R, Herweijer TJ. Height, sitting height and leg length in patients with hypophosphataemic rickets. Acta Paediatr Scand. 1984 Mar;73(2):181-4. doi: 10.1111/j.1651-2227.1984.tb09925.x. PMID 6331056
- [Result] Beccia F, Naso O, Mastrostefano MP. [Indications and limitations of the use of diazepam during labor]. Acta Anaesthesiol. 1968;19:Suppl 9:444+. No abstract available. Italian. PMID 5757628
- [Result] Mietkiewski K, Warchol J, Wojtowicz M, Kosowicz J. [Histological and histochemical examinations of rudimentary gonads]. Endokrynol Pol. 1968 Jul-Aug;19(4):411-27. No abstract available. Polish. PMID 5700869
- [Result] Bunina TL, Rafalovskaia IIa. [Vascular changes in amyotrophic lateral sclerosis]. Zh Nevropatol Psikhiatr Im S S Korsakova. 1969;69(1):11-7. No abstract available. Russian. PMID 5771480
- [Result] Gallwitz D. Histone methylation. Partial purification of two histone-specific methyltransferases from rat thymus nuclei preferentially methylating histones F2a 1 and F3. Arch Biochem Biophys. 1971 Aug;145(2):650-7. doi: 10.1016/s0003-9861(71)80025-5. No abstract available. PMID 5125211
- [Result] Laabs BH, Lohmann K, Vollstedt EJ, Reinberger T, Nuxoll LM, Kilic-Berkmen G, Perlmutter JS, Loens S, Cruchaga C, Franke A, Dobricic V, Hinrichs F, Grozinger A, Altenmuller E, Bellows S, Boesch S, Bressman SB, Duque KR, Espay AJ, Ferbert A, Feuerstein JS, Frank S, Gasser T, Haslinger B, Jech R, Kaiser F, Kamm C, Kollewe K, Kuhn AA, LeDoux MS, Lohmann E, Mahajan A, Munchau A, Multhaupt-Buell T, Pantelyat A, Pirio Richardson SE, Raymond D, Reich SG, Saunders Pullman R, Schormair B, Sharma N, Sichani AH, Simonyan K, Volkmann J, Wagle Shukla A, Winkelmann J, Wright LJ, Zech M, Zeuner KE, Zittel S, Kasten M, Sun YV, Baumer T, Bruggemann N, Ozelius LJ, Jinnah HA, Klein C, Konig IR. Genetic Risk Factors in Isolated Dystonia Escape Genome-Wide Association Studies. Mov Disord. 2024 Nov;39(11):2110-2116. doi: 10.1002/mds.29968. Epub 2024 Sep 17. PMID 39287592
- [Result] Schill J, Simonyan K, Corsten M, Mathys C, Thiel C, Witt K. Graph-theoretical insights into the effects of aging on the speech production network. Cereb Cortex. 2023 Feb 20;33(5):2162-2173. doi: 10.1093/cercor/bhac198. PMID 35584784
- [Result] Schill J, Zeuner KE, Knutzen A, Todt I, Simonyan K, Witt K. Functional Neural Networks in Writer's Cramp as Determined by Graph-Theoretical Analysis. Front Neurol. 2021 Nov 23;12:744503. doi: 10.3389/fneur.2021.744503. eCollection 2021. PMID 34887826
- [Result] Yao D, O'Flynn LC, Simonyan K. DystoniaBoTXNet: Novel Neural Network Biomarker of Botulinum Toxin Efficacy in Isolated Dystonia. Ann Neurol. 2023 Mar;93(3):460-471. doi: 10.1002/ana.26558. Epub 2022 Dec 14. PMID 36440757
- [Result] Frankford SA, O'Flynn LC, Simonyan K. Sensory processing in the auditory and olfactory domains is normal in laryngeal dystonia. J Neurol. 2023 Apr;270(4):2184-2190. doi: 10.1007/s00415-023-11562-z. Epub 2023 Jan 14. PMID 36640203
- [Result] Battistella G, Simonyan K. Clinical Implications of Dystonia as a Neural Network Disorder. Adv Neurobiol. 2023;31:223-240. doi: 10.1007/978-3-031-26220-3_13. Epub 2023 Jun 21. PMID 37338705
- [Result] Schill J, Simonyan K, Lang S, Mathys C, Thiel C, Witt K. Parkinson's disease speech production network as determined by graph-theoretical network analysis. Netw Neurosci. 2023 Jun 30;7(2):712-730. doi: 10.1162/netn_a_00310. eCollection 2023. PMID 37397896
- See also: NIH grant description — https://reporter.nih.gov/search/P2jjzVFcA0umRIMARNgObA/project-details/9692810